CLINICAL TRIAL: NCT05178979
Title: A Gender Transformative Implementation Strategy With Providers to Improve HIV
Brief Title: A Gender Transformative Implementation Strategy With Providers to Improve HIV Outcomes in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at San Antonio (Other)
Collaborators: Makerere University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: K01MH121663-01A1 (NIH); 1K01MH121663-01A1 (NIH)
Record Dates: First submitted 2021-11-15; First posted 2022-01-05 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: Clinics will be randomly assigned to intervention or control via coin toss. Two cohorts of participants will be recruited from both the intervention arm and control arm. The total number of participants (N=240) represents the patient cohort, for which change in patient HIV engagement outcomes are the primary outcomes of the study. A second cohort of HIV providers will also be recruited (n~80-140) depending on the number of HIV providers per clinic, who will provide secondary outcomes related to change in provider knowledge, attitudes, and skills.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Providers (Experimental): HIV care providers and staff in the intervention arm will receive up to 4 sessions of training. Trained intervention facilitator experienced in health professional trainings will lead the training. The intervention content delivered is aimed to increase HIV providers' knowledge, motivation, skills, and empathy to: 1) equitably deliver ART program guidelines (i.e., quality of care) and 2) provide gender sensitive counseling to address ART patients' gendered barriers to HIV care engagement, increasing patient satisfaction, retention, and ART adherence, and reducing gender disparities in HIV outcomes.
  Interventions: Behavioral: Training for HIV care providers (effect on provider outcomes)
- Intervention Clients (Experimental): In the intervention arm clinics, we will enroll a cohort of people living with HIV receiving HIV treatment at the clinics. While they do not receive a direct intervention, we measure change in their outcomes to assess if the provider training intervention has effects on client outcomes.
  Interventions: Behavioral: Training for HIV care providers (effect on provider outcomes)
- Control Providers (No Intervention): The control arm will receive no training. This cohort is of HIV care providers and staff at clinics receiving no intervention.
- Control Clients (No Intervention): The control arm will receive no training. This cohort is of people living with HIV receiving HIV treatment at the control clinics, receiving no intervention.

INTERVENTIONS:
Behavioral: Training for HIV care providers (effect on provider outcomes) — This training program integrates evidence-based strategies to reduce provider bias, adapted to address gender bias in the context of HIV care in Uganda. The content aims to increase providers' knowledge, motivation, skills, and empathy to equitably deliver Ugandan Ministry of Health ART program guidelines to male and female patients (e.g., increasing awareness of HIV gender disparities, increasing empathy/skills to counsel men and women's gendered barriers to care, promoting shared decision-making). The intervention is delivered in a series of group training sessions with HIV providers.
  Arms: Intervention Clients; Intervention Providers

SUMMARY:
Gender norms embedded in the health-system and broader community shape patient-provider relationships in ways that may undermine the provision of antiretroviral treatment (ART) counseling for men and women in Uganda. This study seeks to develop and evaluate the acceptability, feasibility, and preliminary efficacy of an innovative gender transformative implementation strategy to improve HIV provider capacity for equitable HIV care and ART adherence counseling.

DETAILED DESCRIPTION:
Antiretroviral treatment (ART) is the single most effective clinical intervention in the fight against HIV. However, in Uganda only 56% of people living with HIV were virally suppressed in 2017 with significant disparities between men and women, suggesting problems with implementation. While gender norms are a known driver of HIV disparities in sub-Saharan Africa, and patient-provider relationships are a key factor in HIV care engagement, little research has focused on the role that gender norms have in shaping the equitable provision of treatment and quality of ART counseling. The overall research objective is to develop and pilot test an implementation strategy to increase providers' capacity to provide equitable and gender-tailored treatment and counseling to HIV-infected men and women.

Delivered to HIV providers, this group training integrates a gender transformative approach with adapted evidence-based strategies to reduce biases and increase gender equitable attitudes. The pilot trial will assess the implementation strategy's effectiveness by comparing changes in provider (competence for gender sensitive care) and in patient outcomes (clinic attendance, ART adherence, viral load) between the training intervention and usual care through 12-months.

The implementation strategy will be assessed through a quasi-experimental pre/post design. Clinics will be randomly assigned to either the intervention or control condition. Providers in the intervention condition will receive a series of group training sessions. All participants in the provider cohort will complete interviewer administered questionnaires at baseline, 6-, and 12- month follow-up. In addition to the assessment of the cohort of HIV providers, the study will obtain additional data on the impact of the provider training on patient outcomes. Patient participants will complete an interviewer administered questionnaire at baseline, 6-, and 12- month follow-up, and will provide permission for the study team to review and extract relevant data from their clinic records related to engagement in HIV care. The total N and primary outcomes reflected in the clinicaltrials.gov database reflects the patient cohort (N=240, 120 per treatment arm). Secondary outcomes are obtained from the provider cohort (n=20-35 providers per clinic).

ELIGIBILITY:
Provider Cohort:

Inclusion Criteria:

* HIV care provider at the selected clinics, including HIV medical and clinical officers, nurses, midwives, linkage facilitators, counselors.
* 18 years of age or older
* Fluent in English or Luganda

Patient Cohort:

Inclusion Criteria:

* HIV-infected
* Enrolled in care at the clinic of recruitment
* pre-ART (newly diagnosed) or newly initiated on ART (within 3 months-1 year) or struggling with treatment adherence, defined in two ways: (1) most recent viral load results unsuppressed as assessed through clinic records; (2) or self-reported non-adherence as by the Adult AIDS Clinical Trials Group (AACTG) scale 4-day adherence recall questions. This scale has demonstrated good construct validity in Uganda and strong correlations with viral load;
* 18 years of age or an emancipated minor
* Fluent in Luganda or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn M Sileo, PhD, MPH, Principal Investigator — University of Texas at San Antonio; Rhoda K. Wanyenze, MBChB, MPH, PhD, Principal Investigator — Makerere School of Pubic Health
Locations (2):
- Uganda (2):
  - Luwero Health HCIV, Luwero
  - Namayumba Health HCIV, Namayumba

IPD SHARING:
Plan to Share IPD: Yes
Quantitative data collected in this trial (baseline, follow-up assessments) will be made available, under the following provisions: (1)The data will be fully de-identified; (2) Access to the data will be made available first to researchers and their students at the two collaborating institutions (within 3 years of study completion): The University of Texas at San Antonio and the Makerere University School of Public Health (MakSPH); 3) 5 years after study completion, data will be made available to those requesting access outside of the collaborating institutions. Qualitative data collected as part of this trial will not be made available, as it is difficult to fully de-identify and to interpret without knowledge of the context.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years after study completion for researchers and students within the collaborating institutions and 5 years after study completion for those outside of the collaborating institutions upon request
Access Criteria: Upon request from the PI

REFERENCES:
- [Derived] Sileo KM, Wanyenze RK, Anecho A, Luttinen RL, Weston K, Mukasa B, Mukama SC, Vermund SH, Dworkin SL, Dovidio JF, Taylor BS, Kershaw TS. Acceptability, feasibility, and factors affecting implementation of a gender-sensitivity training for HIV providers and staff in Uganda: a mixed methods, quasi-experimental controlled pilot trial. BMC Public Health. 2025 May 24;25(1):1925. doi: 10.1186/s12889-025-23008-4. PMID 40413446
- [Derived] Sileo KM, Wanyenze RK, Anecho A, Luttinen R, Semei C, Mukasa B, Musoke W, Vermund SH, Dworkin SL, Dovidio JF, Taylor BS, Kershaw TS. Protocol for the pilot quasi-experimental controlled trial of a gender-responsive implementation strategy with providers to improve HIV outcomes in Uganda. Pilot Feasibility Stud. 2022 Dec 23;8(1):264. doi: 10.1186/s40814-022-01202-0. PMID 36564795

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Providers: Intervention arm providers receiving the training.
  The intervention arm will receive 4 sessions of training. Trained intervention facilitator experienced in health professional trainings will lead the training. The intervention content delivered is aimed to increase HIV providers' knowledge, motivation, skills, and empathy to: 1) equitably deliver ART program guidelines (i.e., quality of care) and 2) provide gender sensitive counseling to address ART patients' gendered barriers to HIV care engagement, increasing patient satisfaction, retention, and ART adherence, and reducing gender disparities in HIV outcomes.
  Training: This training program integrates evidence-based strategies to reduce provider bias, adapted to address gender bias in the context of HIV care in Uganda. The content aims to increase providers' knowledge, motivation, skills, and empathy to equitably deliver Ugandan Ministry of Health ART program guidelines to male and female patients (e.g., increasing awareness of HIV gender disparities, increasing empathy/skills to counsel men and women's gendered barriers to care, promoting shared decision-making). The intervention is delivered in a series of group training sessions with HIV providers.
- Intervention Clients: Clients receiving HIV care at the intervention arm clinics.
- Control Providers: HIV care providers and staff at the control arm clinics.
- Control Clients: Clients receiving HIV care at the control arm clinics.
Period: Overall Study
Arm/Group | Intervention Providers | Intervention Clients | Control Providers | Control Clients
Started | 61 | 119 | 83 | 119
6-month Follow-up | 60 | 97 | 78 | 91
Completed (12-month follow-up) | 60 | 105 | 80 | 108
Not Completed | 1 | 14 | 3 | 11
Not completed — Death | 0 | 5 | 0 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 8 | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Intervention Providers: HIV care providers and staff receiving the training intervention.
  The intervention arm will receive 4 sessions of training. Trained intervention facilitator experienced in health professional trainings will lead the training. The intervention content delivered is aimed to increase HIV providers' knowledge, motivation, skills, and empathy to: 1) equitably deliver ART program guidelines (i.e., quality of care) and 2) provide gender sensitive counseling to address ART patients' gendered barriers to HIV care engagement, increasing patient satisfaction, retention, and ART adherence, and reducing gender disparities in HIV outcomes.
  Training: This training program integrates evidence-based strategies to reduce provider bias, adapted to address gender bias in the context of HIV care in Uganda. The content aims to increase providers' knowledge, motivation, skills, and empathy to equitably deliver Ugandan Ministry of Health ART program guidelines to male and female patients (e.g., increasing awareness of HIV gender disparities, increasing empathy/skills to counsel men and women's gendered barriers to care, promoting shared decision-making). The intervention is delivered in a series of group training sessions with HIV providers.
- Intervention Clients: Clients receiving HIV care in the intervention arm clinics.
- Control Providers: HIV care providers and staff in the control arm clinics (no intervention).
- Control Clients: Clients receiving HIV care in the control arm clinics (no intervention).
- Total: Total of all reporting groups
Arm/Group | Intervention Providers | Intervention Clients | Control Providers | Control Clients | Total
Number analyzed (Participants) | 61 | 119 | 83 | 119 | 382
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.80 (10.8) | 38.36 (11.66) | 34.9 (10.7) | 39.58 (11.05) | 36.16 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 60 | 59 | 59 | 223
  Male | 16 | 59 | 24 | 60 | 159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 61 | 119 | 83 | 119 | 382
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 61 | 119 | 83 | 119 | 382

OUTCOME MEASURES:

1. Primary Outcome: Change in Proportion of Missed Antiretroviral (ARV) Doses From Baseline Among Clients
Description: AACTG Adherence Instruments, self-reported questionnaire on medication adherence from the Adult AIDS Clinical Trials Group (AACTG); operationalized as a proportion of total missed doses (missed doses/total doses) (continuous measure, range =0.0-1.0)
Time Frame: Baseline, 6-months, and 12-months
Population: The client cohort only is analyzed for this outcome
Measure: Mean (Standard Deviation); unit: percentage of total missed ARV doses
Groups:
- Intervention Clients: Clients receiving HIV care at the intervention clinics.
  The intervention arm will receive 4 sessions of training. Trained intervention facilitator experienced in health professional trainings will lead the training. The intervention content delivered is aimed to increase HIV providers' knowledge, motivation, skills, and empathy to: 1) equitably deliver ART program guidelines (i.e., quality of care) and 2) provide gender sensitive counseling to address ART patients' gendered barriers to HIV care engagement, increasing patient satisfaction, retention, and ART adherence, and reducing gender disparities in HIV outcomes.
  Training: This training program integrates evidence-based strategies to reduce provider bias, adapted to address gender bias in the context of HIV care in Uganda. The content aims to increase providers' knowledge, motivation, skills, and empathy to equitably deliver Ugandan Ministry of Health ART program guidelines to male and female patients (e.g., increasing awareness of HIV gender disparities, increasing empathy/skills to counsel men and women's gendered barriers to care, promoting shared decision-making). The intervention is delivered in a series of group training sessions with HIV providers.
- Control Clients: Clients receiving HIV care at the control clinics.
Arm/Group | Intervention Clients | Control Clients
Number analyzed (Participants) | 105 | 108
percentage of total missed ARV doses
  Baseline | 90.14 (19.51) | 91.68 (22.40)
  6-months | 95.64 (14.35) | 96.73 (13.33)
  12-months | 95.45 (19.51) | 100.00 (0.00)
Statistical Analysis 1: Comparison: Control Clients; Test type: Superiority; p = 0.38, Regression, Linear — Models control for clinic, gender, lifetime experience of intimate partner violence (IPV) and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Wald Chi-Square = 1.94 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Clients; Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Test type: Superiority; p = 0.84, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; Models control for clinic, gender, lifetime experience of intimate partner violence (IPV) and are adjusted for multiple time points; unstandardized beta = 0.93, Standard Error of Mean 4.63
Statistical Analysis 3: Comparison: Control Clients; Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Test type: Superiority; p = 0.50, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; [statistical method as in outcome 1, analysis 2]; unstandardized beta = -2.62, Standard Error of Mean 3.87

2. Primary Outcome: Change in Clinic Visit Adherence From Baseline Among Patients (Retention in Care)
Description: Proportion of kept visits/scheduled visits (kept + missed visits) (continuous measure, range =0.0-1.0)
Time Frame: Baseline, 6-months, and 12-months
Population: The client cohort only is analyzed for this outcome
Measure: Mean (Standard Deviation); unit: percentage of total missed visits
Groups:
- Intervention Clients: Clients receiving HIV care at the intervention clinics.
  The intervention arm will receive 4 sessions of training. Trained intervention facilitator experienced in health professional trainings will lead the training. The intervention content delivered is aimed to increase HIV providers' knowledge, motivation, skills, and empathy to: 1) equitably deliver ART program guidelines (i.e., quality of care) and 2) provide gender sensitive counseling to address ART patients' gendered barriers to HIV care engagement, increasing patient satisfaction, retention, and ART adherence, and reducing gender disparities in HIV outcomes.
  Training: This training program integrates evidence-based strategies to reduce provider bias, adapted to address gender bias in the context of HIV care in Uganda. The content aims to increase providers' knowledge, motivation, skills, and empathy to equitably deliver Ugandan Ministry of Health ART program guidelines to male and female patients (e.g., increasing awareness of HIV gender disparities, increasing empathy/skills to counsel men and women's gendered barriers to care, promoting shared decision-making). The intervention is delivered in a series of group training sessions with HIV providers.
  Each study arm has 2 cohorts: HIV care providers/staff and HIV care clients
Arm/Group | Intervention Clients | Control Clients
Number analyzed (Participants) | 105 | 108
percentage of total missed visits
  Baseline | 0.96 (0.11) | 0.95 (0.12)
  6-months | 0.99 (0.06) | 0.98 (0.08)
  12-months | 0.99 (0.07) | 1.00 (0.00)
Statistical Analysis 1: Comparison: Control Clients; Test type: Superiority; p = 0.37, Regression, Linear — Models control for clinic and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Wald Chi-square = 2.00 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Clients; Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Test type: Superiority; p = 0.18, Regression, Linear — P-value is adjusted for clinic; this value is the 6-month follow-up; Model controls for clinic; unstandardized beta = -0.02, Standard Error of Mean 0.01
Statistical Analysis 3: Comparison: Control Clients; Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Test type: Superiority; p = 0.19, Regression, Linear — P-value is adjusted for clinic; this value is the 12-month follow-up; Model controls for clinic; unstandardized beta = -0.03, Standard Error of Mean 0.02 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints

3. Primary Outcome: Change in Competence for Gender-sensitive Care From Baseline Among Providers
Description: Adapted from the Nijmegen Gender Awareness in Medicine Scale (N-GAMS); collected from provider cohort; 9 items, total possible score using mean scoring: 1-5 (high score = better outcome)
Time Frame: Baseline, 6-months, and 12-months
Population: The provider cohort only is analyzed for this outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Providers: HIV care providers/staff at the intervention clinics.
  The intervention arm will receive 4 sessions of training. Trained intervention facilitator experienced in health professional trainings will lead the training. The intervention content delivered is aimed to increase HIV providers' knowledge, motivation, skills, and empathy to: 1) equitably deliver ART program guidelines (i.e., quality of care) and 2) provide gender sensitive counseling to address ART patients' gendered barriers to HIV care engagement, increasing patient satisfaction, retention, and ART adherence, and reducing gender disparities in HIV outcomes.
  Training: This training program integrates evidence-based strategies to reduce provider bias, adapted to address gender bias in the context of HIV care in Uganda. The content aims to increase providers' knowledge, motivation, skills, and empathy to equitably deliver Ugandan Ministry of Health ART program guidelines to male and female patients (e.g., increasing awareness of HIV gender disparities, increasing empathy/skills to counsel men and women's gendered barriers to care, promoting shared decision-making). The intervention is delivered in a series of group training sessions with HIV providers.
  Each study arm has 2 cohorts: HIV care providers/staff and HIV care clients
- Control Providers: HIV care providers/staff at the control clinics.
Arm/Group | Intervention Providers | Control Providers
Number analyzed (Participants) | 60 | 78
score on a scale
  Baseline | 3.78 (0.40) | 3.55 (0.24)
  6-month | 3.95 (0.35) | 3.48 (0.25)
  12-month | 3.82 (0.31) | 3.61 (0.31)
Statistical Analysis 1: Comparison: Control Providers; Test type: Superiority; p = 0.004, Regression, Linear — Models control for clinic, cadre, and gender and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Wald Chi-square = 10.84 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Providers; Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; Models control for clinic, cadre, and gender and are adjusted for multiple time points; unstandardized beta = 0.24, Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Control Providers; Test type: Superiority; p = 0.86, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; Models control for clinic, cadre, and gender and are adjusted for multiple time points; unstandardized beta = -0.02, Standard Error of Mean 0.09

4. Secondary Outcome: Change in Self-efficacy for Client-centered Communication From Baseline Among Providers
Description: An adapted version of the Self-Efficacy Questionnaire (SE-12) for Provider Communication was used to assess communication self-efficacy, adapted to be gender specific. 5 items. Total possible score using mean scoring: 0-4 (high score = better outcome)
Time Frame: Baseline, 6-months, and 12-months
Population: The provider cohort only is analyzed for this outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Providers: HIV care providers/staff at the intervention clinics.
  The intervention arm will receive 4 sessions of training. Trained intervention facilitator experienced in health professional trainings will lead the training. The intervention content delivered is aimed to increase HIV providers' knowledge, motivation, skills, and empathy to: 1) equitably deliver ART program guidelines (i.e., quality of care) and 2) provide gender sensitive counseling to address ART patients' gendered barriers to HIV care engagement, increasing patient satisfaction, retention, and ART adherence, and reducing gender disparities in HIV outcomes.
  Training: This training program integrates evidence-based strategies to reduce provider bias, adapted to address gender bias in the context of HIV care in Uganda. The content aims to increase providers' knowledge, motivation, skills, and empathy to equitably deliver Ugandan Ministry of Health ART program guidelines to male and female patients (e.g., increasing awareness of HIV gender disparities, increasing empathy/skills to counsel men and women's gendered barriers to care, promoting shared decision-making). The intervention is delivered in a series of group training sessions with HIV providers.
Arm/Group | Intervention Providers | Control Providers
Number analyzed (Participants) | 60 | 78
score on a scale
  Baseline | 3.08 (0.75) | 3.15 (0.40)
  6-month | 3.24 (0.54) | 3.26 (0.43)
  12-month | 2.98 (0.53) | 3.28 (0.49)
Statistical Analysis 1: Comparison: Control Providers; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Wald Chi-square = 21.42 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Providers; update; Test type: Superiority; p = 0.81, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; Models control for clinic, cadre, and gender and are adjusted for multiple time points; unstandardized beta = 0.04, Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Control Providers; update; Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; Models control for clinic, cadre, and gender and are adjusted for multiple time points; unstandardized beta = -0.22, Standard Error of Mean 0.07

5. Secondary Outcome: Change in Empathy Towards Clients From Baseline Among Providers
Description: Provider empathy for clients' experiences was measured from an adapted version of the Jefferson Scale of Physician Empathy, which has been adapted for HIV care previously. 9 items, total possible score using mean scoring: 1-5 (high score = better outcome)
Time Frame: Baseline, 6-months, and 12-months
Population: The provider cohort only is analyzed for this outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Providers | Control Providers
Number analyzed (Participants) | 60 | 78
score on a scale
  Baseline | 3.77 (0.38) | 3.62 (0.38)
  6-month | 3.86 (0.45) | 3.54 (0.32)
  12-month | 3.91 (0.30) | 3.63 (0.44)
Statistical Analysis 1: Comparison: Control Providers; Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 3, analysis 1]; Wald Chi-square = 150.43 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Providers; Test type: Superiority; p = 0.002, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; unstandardized beta = 0.17, Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Control Providers; Test type: Superiority; p = 0.03, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; unstandardized beta = 0.13, Standard Error of Mean 0.06

6. Secondary Outcome: Change in the Use of Emotional Regulation and Stress Reduction Techniques From Baseline Among Providers
Description: Providers' use of emotional regulation and stress reduction techniques, such as breathing exercises, sense soothing, tension release, attention shifting, and positive reframing, were measured through items adapted from the Mindful Self-Care Scale (MSCS) and the Brief COPE. 7-items, total possible score using mean scoring: 0-4 (high score = better outcome)
Time Frame: Baseline, 6-months, and 12-months
Population: The provider cohort only is analyzed for this outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Providers | Control Providers
Number analyzed (Participants) | 60 | 78
score on a scale
  Baseline | 1.64 (0.91) | 1.99 (0.62)
  6-month | 1.93 (0.80) | 1.86 (0.75)
  12-month | 2.03 (0.97) | 2.06 (0.81)
Statistical Analysis 1: Comparison: Control Providers; Test type: Superiority; p = 0.01, Regression, Linear — [p-value comment as in outcome 3, analysis 1]; Wald Chi-square = 8.72 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Providers; Test type: Superiority; p = 0.15, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; Models control for clinic, cadre, and gender and are adjusted for multiple time points; unstandardized beta = 0.42, Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Control Providers; Test type: Superiority; p = 0.008, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; Models control for clinic, cadre, and gender and are adjusted for multiple time points; unstandardized beta = 0.32, Standard Error of Mean 0.12

7. Secondary Outcome: Change in Perceived Quality of Communication From HIV Providers From Baseline Among Clients
Description: Patient's perceptions of the quality of communication with their HIV care providers was measured through two scales that were combined for a total score continuous score. Wilson et al. was developed for HIV populations, including items measuring the perceived quality of general health communication from HIV care providers, asking patients to rate the quality of their HIV care providers in communicating general health information and in providing HIV specific information. In addition, patients' perceived quality of provider communication specific to ART adherence was be measured from items adapted from Schneider and colleagues. 14 items, total possible score using mean scoring: 0-4 (high score = better outcome)
Time Frame: Baseline, 6-months, and 12-months
Population: The client cohort only is analyzed for this outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Clients | Control Clients
Number analyzed (Participants) | 105 | 108
score on a scale
  Baseline | 2.33 (0.86) | 2.25 (0.69)
  6-month | 2.53 (1.04) | 2.32 (0.62)
  12-month | 2.14 (0.87) | 2.88 (0.43)
Statistical Analysis 1: Comparison: Control Clients; Test type: Superiority; p < 0.001, Regression, Linear — Models control for clinic and income and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Wald Chi-square = 172.52 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Clients; Test type: Superiority; p = 0.68, Regression, Linear — P-value is adjusted for multiple comparisons; this value is the 6-month follow-up; Models control for clinic and income and are adjusted for multiple time points; unstandardized beta = 0.14, Standard Error of Mean 0.34
Statistical Analysis 3: Comparison: Control Clients; Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; Models control for clinic and income and are adjusted for multiple time points; unstandardized beta = -0.83, Standard Error of Mean 0.24

8. Secondary Outcome: Change in Perceived Level of Participatory Decision-making Related to HIV Care From Baseline Among Clients
Description: Participatory decision-making style of HIV care providers, or how active of a role patients perceive they have in their health care decisions, was measured with Kaplan's 7-item scale. Total possible score using mean scoring: 0-4 (high score = better outcome)
Time Frame: Baseline, 6-months, and 12-months
Population: The client cohort only is analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Clients | Control Clients
Number analyzed (Participants) | 105 | 108
score on a scale
  Baseline | 1.86 (1.04) | 2.19 (0.97)
  6-month | 2.11 (0.90) | 2.69 (0.79)
  12-month | 2.52 (0.93) | 2.75 (0.39)
Statistical Analysis 1: Comparison: Control Clients; Test type: Superiority — Models control for clinic, income, years living with HIV and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; p < 0.001, Regression, Linear; Wald Chi-square = 25.27 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Clients; Test type: Superiority; p = 0.10, Regression, Linear — P-value is adjusted for multiple comparisons; this value is the 6-month follow-up; Models control for clinic, income, years living with HIV and are adjusted for multiple time points; unstandardized beta = -0.26, Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Control Clients; Test type: Superiority; p = 0.54, Regression, Linear — P-value is adjusted for multiple comparisons; this value is the 12-month follow-up; Models control for clinic, income, years living with HIV and are adjusted for multiple time points; unstandardized beta = 0.08, Standard Error of Mean 0.14

9. Secondary Outcome: Change in Satisfaction With HIV Care From Baseline Among Clients
Description: The GHAA Consumer Satisfaction Survey measures overall satisfaction with care; we adapted these items to focus specifically on HIV care to measure patient satisfaction with HIV care. 6 items, total possible score using mean scoring: 0-4 (high score = better outcome)
Time Frame: Baseline, 6-months, and 12-months
Population: The client cohort only is analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Clients | Control Clients
Number analyzed (Participants) | 105 | 108
score on a scale
  Baseline | 3.38 (0.55) | 3.26 (0.35)
  6-month | 3.29 (0.60) | 3.19 (0.40)
  12-month | 3.09 (0.59) | 3.27 (0.33)
Statistical Analysis 1: Comparison: Control Clients; Test type: Superiority — Models control for clinic, gender, AUDIT score and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; p < 0.001, Regression, Linear — Models control for clinic, gender, AUDIT score and are adjusted for multiple time points; Wald Chi-square = 36.04 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Clients; Test type: Superiority; p = 0.97, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; Models control for clinic, gender, AUDIT score and are adjusted for multiple time points; unstandardized beta = -0.00, Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Control Clients; Test type: Superiority; p < 0.001, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; Models control for clinic, gender, AUDIT score and are adjusted for multiple time points; unstandardized beta = -0.29, Standard Error of Mean 0.07

10. Secondary Outcome: Change in Total HIV Stigma Score Among Clients
Description: HIV stigma was measured using Earnshaw's HIV stigma framework scale , which measures anticipated (the degree of HIV stigma one expects to encounter from others), enacted (the degree of HIV stigma one has encountered from others), and internalized HIV stigma (the degree to which one internalized negative beliefs about people living with HIV about themselves). This outcome reports the mean for the entire scale. 21 items, total possible score using mean scoring: 0-4 (high score = worse outcome).
Time Frame: Baseline, 6-months, and 12-months
Population: The client cohort only is analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Clients | Control Clients
Number analyzed (Participants) | 105 | 108
score on a scale
  Baseline | 0.60 (0.65) | 0.60 (0.57)
  6-month | 0.59 (0.66) | 0.58 (0.55)
  12-month | 0.45 (0.64) | 0.71 (0.50)
Statistical Analysis 1: Comparison: Control Clients; Test type: Superiority; p = 0.01, Regression, Linear — Models control for clinic, gender, years living with HIV, AUDIT score and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Wald Chi-square = 9.46 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Clients; Test type: Superiority; p = 0.81, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; Models control for clinic, gender, years living with HIV, AUDIT score and are adjusted for multiple time points; unstandardized beta = 0.03, Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Control Clients; Test type: Superiority; p = 0.04, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; Models control for clinic, gender, years living with HIV, AUDIT score and are adjusted for multiple time points; unstandardized beta = -0.25, Standard Error of Mean 0.13

11. Secondary Outcome: Change in Anticipated HIV Stigma Among Clients
Description: HIV stigma was measured using Earnshaw's HIV stigma framework scale , which measures anticipated (the degree of HIV stigma one expects to encounter from others), enacted (the degree of HIV stigma one has encountered from others), and internalized HIV stigma (the degree to which one internalized negative beliefs about people living with HIV about themselves). This outcome reports the mean for the anticipated scale. 7 items, total possible score using mean scoring: 0-4 (high score = worse outcome).
Time Frame: Baseline, 6-months, and 12-months
Population: The client cohort only is analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Clients | Control Clients
Number analyzed (Participants) | 105 | 108
score on a scale
  Baseline | 0.79 (0.89) | 0.67 (0.89)
  6-month | 0.80 (0.88) | 0.57 (0.73)
  12-month | 0.59 (0.88) | 0.90 (0.63)
Statistical Analysis 1: Comparison: Control Clients; Test type: Superiority; p < 0.001, Regression, Linear — Models control for clinic, gender, years living with HIV and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Wald Chi-square = 14.77 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Clients; Test type: Superiority; p = 0.45, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; Models control for clinic, gender, years living with HIV and are adjusted for multiple time points; unstandardized beta = 0.12, Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Control Clients; Test type: Superiority; p = 0.02, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; Models control for clinic, gender, years living with HIV and are adjusted for multiple time points; unstandardized beta = -0.43, Standard Error of Mean 0.18

12. Secondary Outcome: Change in Enacted HIV Stigma Among Clients
Description: HIV stigma was measured using Earnshaw's HIV stigma framework scale , which measures anticipated (the degree of HIV stigma one expects to encounter from others), enacted (the degree of HIV stigma one has encountered from others), and internalized HIV stigma (the degree to which one internalized negative beliefs about people living with HIV about themselves). This outcome reports the mean for the enacted scale. 7 items, total possible score using mean scoring: 0-4 (high score = worse outcome).
Time Frame: Baseline, 6-months, and 12-months
Population: The client cohort only is analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Clients: Clients receiving HIV care at the intervention clinics.
Arm/Group | Intervention Clients | Control Clients
Number analyzed (Participants) | 105 | 108
score on a scale
  Baseline | 0.21 (0.52) | 0.14 (0.43)
  6-month | 0.16 (0.46) | 0.14 (0.42)
  12-month | 0.12 (0.39) | 0.17 (0.47)
Statistical Analysis 1: Comparison: Control Clients; Test type: Superiority; p = 0.004, Regression, Linear — Models control for clinic, AUDIT score, food insecurity and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Wald Chi-square = 11.06 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Clients; Test type: Superiority; p = 0.35, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; Models control for clinic, AUDIT score, food insecurity and are adjusted for multiple time points; unstandardized beta = -0.06, Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Control Clients; Test type: Superiority; p = 0.04, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; Models control for clinic, AUDIT score, food insecurity and are adjusted for multiple time points; unstandardized beta = -0.13, Standard Error of Mean 0.06

13. Secondary Outcome: Change in Internalized HIV Stigma Among Clients
Description: HIV stigma was measured using Earnshaw's HIV stigma framework scale , which measures anticipated (the degree of HIV stigma one expects to encounter from others), enacted (the degree of HIV stigma one has encountered from others), and internalized HIV stigma (the degree to which one internalized negative beliefs about people living with HIV about themselves). This outcome reports the mean for the internalized scale. 7 items, total possible score using mean scoring: 0-4 (high score = worse outcome).
Time Frame: Baseline, 6-months, and 12-months
Population: The client cohort only is analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Clients | Control Clients
Number analyzed (Participants) | 105 | 108
score on a scale
  Baseline | 0.78 (1.13) | 0.99 (0.85)
  6-month | 0.82 (1.14) | 1.01 (0.95)
  12-month | 0.62 (0.99) | 1.04 (0.61)
Statistical Analysis 1: Comparison: Control Clients; Test type: Superiority; p = 0.24, Regression, Linear — Models control for clinic, gender, years living with HIV, travel time to clinic and are adjusted for multiple time points. Models run using generalized estimating equations (GEE) to account for dependence in repeated, clustered data; Wald Chi-square = 2.84 — Wald Chi-Square tests the overall arm*time intervention effect across the timepoints
Statistical Analysis 2: Comparison: Control Clients; Test type: Superiority; p = 0.92, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 6-month follow-up; Models control for clinic, gender, years living with HIV, travel time to clinic and are adjusted for multiple time points; unstandardized beta = 0.02, Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Control Clients; Test type: Superiority; p = 0.21, Regression, Linear — P-value is adjusted for multiple comparisons; this value is for the 12-month follow-up; [statistical method as in outcome 13, analysis 2]; unstandardized beta = -0.21, Standard Error of Mean 0.16

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Control Providers: HIV care providers and staff at the control clinics (no intervention).
- Control Clients: Clients receiving HIV care at the control clinics (no intervention).
Arm/Group | Intervention Providers | Intervention Clients | Control Providers | Control Clients
All-Cause Mortality (participants affected / at risk) | 0/61 | 5/119 | 0/83 | 3/119
Serious Adverse Events (participants affected / at risk) | 0/61 | 1/119 | 0/83 | 0/119
Other Adverse Events (participants affected / at risk) | 0/61 | 0/119 | 0/83 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Providers (N=61) | Intervention Clients (N=119) | Control Providers (N=83) | Control Clients (N=119)
Mental health (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — 1 participant hospitalized due to mental health problems

LIMITATIONS AND CAVEATS:
This study is a pilot trial. Therefore, the results reported are exploratory because they are underpowered. A full-scale efficacy trial is needed to replicate these results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT05178979/Prot_SAP_000.pdf